CLINICAL TRIAL: NCT04188964
Title: A Phase 1/2, Open-label, Multicenter, Non-randomized Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of Burosumab in Pediatric Patients From Birth to Less Than 1 Year of Age With X-linked Hypophosphatemia (XLH)
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of Burosumab in Patients Less Than 1 Year of Age
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Pharmaceutical Development Ltd (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUR-CL207
Record Dates: First submitted 2019-11-25; First posted 2019-12-06 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: X-linked Hypophosphatemia (XLH)
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Pediatric subjects > = 6 months to < 12 months will receive a starting dose of 0.4mg/kg administered subcutaneously (SC) every 2 weeks (Q2W) for 48 weeks with the option of the dose to be increased to 0.8mg/kg upon recommendation of the Data Safety Management Board (DSMB). The dose can be either increased up to a maximum of 2 mg/kg or decreased to 0.2 mg/kg depending on serum phosphate response. Upon recommendation of the DSMB subjects < 6 months can then start at 0.4mg/kg starting dose administered subcutaneously (SC) every 2 weeks (Q2W) for 48 weeks with the option to be increased to 0.8mg/kg upon recommendation of the DSMB and can be either increased up to a maximum of 2 mg/kg or decreased to 0.2 mg/kg depending on serum phosphate response.
  Interventions: Drug: Burosumab

INTERVENTIONS:
Drug: Burosumab — Burosumab is a sterile clear colourless to slightly yellow and preservative free solution supplied in single use 5ml vials containing 1 mL of Burosumab at a concentration of 10mg/mL,20 mg/mL or 30mg/mL, administered by SC injections every 2 weeks.
  Other Names: KRN23; Crysvita

SUMMARY:
A Phase 1/2, Open-label, Multicenter, Non-randomized Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of Burosumab in Paediatric Patients from Birth to Less than 1 Year of Age with X-linked Hypophosphatemia (XLH)

DETAILED DESCRIPTION:
BUR-CL207 is a multicenter, open-label, non-randomized Phase 1/2 study in pediatric patients with XLH initiating treatment with burosumab at <12 months of age. The study includes a total treatment period of up to 48 weeks across 3 cohorts. Subjects will be enrolled in 2 age subgroups: (1) ≥6 months to <12 months of age, and (2) <6 months of age at initiation of burosumab treatment. Cohorts will aim to include 3 subjects per cohort depending on the starting dose of burosumab and relative response of patients to treatment as assessed by serum phosphate levels and by the treating physician (Investigator). Cohorts will commence in a staggered manner starting with Cohort 1, followed by Cohorts 2 and 3, which may start in parallel after an adequate observation period (4 weeks) in Cohort 1 and with approval from the Sponsor's Medical Monitor and the DSMB. The cohorts are defined as follows:

* Cohort 1: pediatric subjects with XLH and hypophosphatemia (serum phosphate below the age-adjusted lower limit of normal [LLN]), and age from ≥6 months to <12 months of age at initiating treatment with burosumab with starting dose of 0.4 mg/kg.
* Cohort 2: pediatric subjects with XLH and hypophosphatemia (serum phosphate below the age-adjusted LLN), and age from ≥6 months to <12 months of age at initiating treatment with burosumab with a starting dose of 0.8 mg/kg (upon Data Safety Monitoring Board [DSMB] confirmation).
* Cohort 3: pediatric subjects with XLH and hypophosphatemia (serum phosphate below the age-adjusted LLN), and <6 months of age at initiating treatment with burosumab with a starting dose of 0.4 mg/kg (upon DSMB confirmation). Following enrollment of the first 3 or 4 subjects in Cohort 3, an interim population PK/PD evaluation may be performed to determine whether the starting dose for the cohort can be increased to 0.8 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female pediatric subjects, aged <12 months at burosumab treatment initiation.
2. Pediatric subjects with PHEX mutation or variant of uncertain significance in either the subject or a directly related family member with appropriate X-linked inheritance.
3. Presenting serum phosphate levels below the age-specific LLN at Screening.
4. A legally authorized representative has provided written informed consent prior to any research-related procedures.
5. A legally authorized representative must, in the opinion of the Investigator, be willing and able to complete all aspects of the study, adhere to the study visit schedule, and comply with the assessments required by the study protocol, including providing access to prior medical records for the collection of historical growth, biochemical, and radiographic data and disease history.

Exclusion Criteria:

1. The pediatric subject's legally authorized representative is unwilling or unable to stop the subject's treatment with oral phosphate and/or pharmacologic vitamin D metabolite or analogue (e.g. calcitriol, alfacalcidol) for at least 1 week before planned treatment start and for the duration of the study.
2. Preterm pediatric patients (defined as born before 37 weeks of pregnancy) with a chronological age of <6 months. Enrolment of preterm pediatric patients with a chronological age ≥6 months must be confirmed by the Study Medical Monitor before study entry.
3. Impairment of renal function measured as serum creatinine above the age-adjusted normal range and estimated GFR (calculated using the Bedside Schwartz equation) below the age-adjusted normal range.
4. Presence of nephrocalcinosis on renal ultrasound.
5. Hypocalcemia or hypercalcemia, defined as serum calcium levels outside the age-adjusted normal limits.
6. Presence of a concurrent disease or condition that would interfere with study participation or affect subject safety.
7. Predisposition to infection or known immunodeficiency.
8. Severe dermatological conditions over the available injection sites.
9. Use of any investigational product or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
10. Metabolic bone disease, nutritional rickets and/or osteopenia of other origin than XLH at Screening and/or Baseline.
11. Serum levels of 25-hydroxyvitamin D (25(OH)D) below the LLN that are clinically significant in the opinion of the Investigator.
12. Evidence of any hyperparathyroidism not associated with XLH as determined by the Investigator.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of Burosumab in paediatric subjects with X-linked Hypophosphatemia (XLH) starting treatment below 12 months of age | From Baseline to scheduled time points (measured throughout the study up to Week 48).
  Incidence, frequency, and severity of adverse events (AEs) and serious AEs (SAEs), including clinically significant changes in laboratory, physical examinations, vital signs, ECGs and imaging assessments

SECONDARY OUTCOMES:
To characterize the pharmacokinetics (PK) of Burosumab following subcutaneous (SC) injection in paediatric subjects with XLH below 12 months of age. | Measured throughout the study up to Week 48
  Burosumab serum concentrations and PK parameters, including apparent clearance (CL/F), apparent volume of distribution (V/F), area under the serum concentration-time curve (AUC), maximum serum drug concentration (Cmax) and other parameters, as appropriate.
To characterize the effect of Burosumab on serum phosphate and 1,25-dihydroxyvitamin D (1,25[OH]2D) in paediatric subjects with XLH starting treatment below 12 months of age | Change from Baseline at Week 20, 26, 32, 40 and 48
  Changes in serum phosphate and 1,25-dihydroxyvitamin D (1,25[OH]2D)
To assess the clinical effects of Burosumab on growth and prevention and/or healing of rickets and skeletal deformities | Baseline and Week 48
  Change in serum alkaline phosphatase (ALP).
To assess the clinical effects of Burosumab on growth and prevention and/or healing of rickets and skeletal deformities | At week 48
  Appearance in radiographic appearance of rickets severity as assessed by the Radiograph Global Impression of Change (RGI-C) scoring system.
To assess the clinical effects of burosumab on growth and prevention and/or healing of rickets and skeletal deformities | At week 48
  The appearance in rickets severity assessed by total Rickets Severity Score (RSS).
To assess the clinical effects of burosumab on growth and prevention and/or healing of rickets and skeletal deformities | At week 48
  Change in lower extremity skeletal abnormalities, including genu varum and genu valgus, as determined by the RGI-C long leg score.
To assess the clinical effects of burosumab on growth and prevention and/or healing of rickets and skeletal deformities | At week 48
  Change in recumbent length in cm, height-for-age z-scores, and percentiles.

CONTACTS AND LOCATIONS:
Locations (9):
- Kepler Universitaetsklinikum GmbH, Linz, Austria
- France (2):
  - Centre de reference des maladies renales rares-Hospices Civils de Lyon-Hopital Femme Mere Enfant, Lyon
  - Hopital Kremlin APHP, Paris
- Ospedale Pediatrico Bambino Gesù, Rome, Italy
- Hospital Virgen del Rocío, Seville, Spain
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (3):
  - Evelina London Children's Hospital - Guy's & St Thomas' NHS Foundation Trust, London
  - Great Ormond Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No